CLINICAL TRIAL: NCT02382276
Title: A Long-term Extension Study for the Phase 3 Study of Nalmefene (339-14-001) in Patients With Alcohol Dependence
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Collaborators: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 339-14-002; JapicCTI-152806 (Other: Japic)
Record Dates: First submitted 2015-02-10; First posted 2015-03-06 (Estimated); Results first posted 2020-07-20 (Actual); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Alcohol Dependence
MeSH Terms: conditions — Alcoholism | interventions — nalmefene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nalmefene hydrochloride 20 mg (Experimental): As-needed; tablets, orally
  Interventions: Drug: Nalmefene hydrochloride

INTERVENTIONS:
Drug: Nalmefene hydrochloride

SUMMARY:
The long-term safety and efficacy of nalmefene hydrochloride at 20 mg in patients with alcohol dependence will be evaluated in a multicenter, open-label, uncontrolled trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have completed Study 339-14-001
* Patients who have signed the informed consent form for Study 339-14-002

Exclusion Criteria:

* The patient has a clinically significant unstable illness (eg, complication of New York Heart Association (NYHA) class III or IV heart failure or angina pectoris, renal function disorder with estimated glomerular filtration rate (eGFR) of < 30 mL/min/1.73 m2, hepatic failure, and neoplastic disorder)
* The patient has a clinically significant abnormal electrocardiogram (ECG) which is inappropriate for the participation in the trial in the opinion of the investigator or subinvestigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 405 (Actual)
Dates: Start 2015-07-13 (Actual); Primary Completion 2017-01-18 (Actual); Study Completion 2017-01-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ono Hiroaki, Mr, Study Director — Otsuka Pharmaceutical Co., Ltd.
Locations (7):
- Japan (7):
  - Chubu, Region
  - Hokkaido, Region
  - Kanto, Region
  - Kinki, Region
  - Kyusyu, Region
  - Tohoku, Region
  - Tyugoku, Region

RESULTS

PARTICIPANT FLOW:
Groups:
- Nalmefene 20 mg in the lead-in Study: Patients who completed the treatment (nalmefene hydrochloride 20 mg) in the lead-in study were eligible for the extension study. In the extension study, all patients were received nalmefene 20 mg tablets, as-needed, orally, 24-week treatment period.
- Nalmefene 10 mg in the lead-in Study: Patients who completed the treatment (nalmefene hydrochloride 10 mg) in the lead-in study were eligible for the extension study. In the extension study, all patients were received nalmefene 20 mg tablets, as-needed, orally, 24-week treatment period.
- Placebo in the lead-in Study: Patients who completed the treatment (placebo) in the lead-in study were eligible for the extension study. In the extension study, all patients were received nalmefene 20 mg tablets, as-needed, orally, 24-week treatment period.
Period: Overall Study
Arm/Group | Nalmefene 20 mg in the lead-in Study | Nalmefene 10 mg in the lead-in Study | Placebo in the lead-in Study
Started | 137 | 94 | 172
Completed | 126 | 84 | 133
Not Completed | 11 | 10 | 39
Not completed — Withdrawal by Subject | 4 | 8 | 5
Not completed — Adverse Event | 7 | 2 | 32
Not completed — Physician Decision | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Safety analysis set, which included all patients who received at least one dose of study medication during the 24-week treatment period in the extension study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Nalmefene 20 mg in the lead-in Study | Nalmefene 10 mg in the lead-in Study | Placebo in the lead-in Study | Total
Number analyzed (Participants) | 137 | 94 | 172 | 403
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 120 | 85 | 154 | 359
  >=65 years | 17 | 9 | 18 | 44
Age, Customized [Mean (Standard Deviation); unit: years] | 50.0 (11.7) | 50.1 (11.0) | 48.5 (11.0) | 49.4 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 19 | 64 | 116
  Male | 104 | 75 | 108 | 287
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Japanese | 137 | 94 | 172 | 403
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 137 | 94 | 172 | 403
Heavy Drinking Days (HDDs) [Mean (Standard Deviation); unit: days/month] — The number of HDDs was defined as the number of days per month [days/month] with alcohol consumption of > 60 g for males and > 40 g for females. Population: Full analysis set, which included all patients from the SS who had data available for HDDs at baseline in the lead-in study and at one or more time-points in the extension study.
  days/month
    number analyzed (Participants) | 137 | 94 | 169 | 400
    (all) | 22.54 (6.70) | 24.38 (5.10) | 22.70 (6.54) | 23.04 (6.32)
Total Alcohol Consumption (TAC) [Mean (Standard Deviation); unit: g/day] — TAC was defined as mean alcohol consumption per day [g/day] over a 1-month period. Population: Full analysis set, which included all patients from the SS who had data available for HDDs at baseline in the lead-in study and at one or more time-points in the extension study.
  g/day
    number analyzed (Participants) | 137 | 94 | 169 | 400
    (all) | 94.10 (34.43) | 94.16 (32.60) | 92.30 (41.03) | 93.35 (36.90)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Time Frame: 24-week treatment period
Population: as for baseline characteristics
Measure: Number; unit: Number of participants
Arm/Group | Nalmefene 20 mg in the lead-in Study | Nalmefene 10 mg in the lead-in Study | Placebo in the lead-in Study
Number analyzed (Participants) | 137 | 94 | 172
Number of participants | 96 | 67 | 141

2. Secondary Outcome: Change in the Number of Heavy Drinking Days (HDDs) From Baseline
Time Frame: Week 24
Population: Full analysis set, which included all patients from the SS who had data available for HDDs at baseline in the lead-in study and at one or more time-points in the extension study.
Measure: Least Squares Mean (Standard Error); unit: days/month
Arm/Group | Nalmefene 20 mg in the lead-in Study | Nalmefene 10 mg in the lead-in Study | Placebo in the lead-in Study
Number analyzed (Participants) | 137 | 94 | 169
days/month | -15.09 (0.77) | -17.15 (0.94) | -16.35 (0.70)

3. Secondary Outcome: Change in Total Alcohol Consumption (TAC) From Baseline
Time Frame: Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: g/day
Arm/Group | Nalmefene 20 mg in the lead-in Study | Nalmefene 10 mg in the lead-in Study | Placebo in the lead-in Study
Number analyzed (Participants) | 137 | 94 | 169
g/day | -53.20 (2.29) | -57.93 (2.77) | -55.77 (2.06)

ADVERSE EVENTS:
Time Frame: 24-week treatment period
Groups:
- Total: Nalmefene 20 mg tablets, as-needed, orally, 24-week treatment period in the extension study
Arm/Group | Total
All-Cause Mortality (participants affected / at risk) | 0/403
Serious Adverse Events (participants affected / at risk) | 3/403
Other Adverse Events (participants affected / at risk) | 209/403
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Total (N=403)
Gastroenteritis (Infections and infestations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Total (N=403)
Abdominal discomfort (Gastrointestinal disorders) | 23
Nausea (Gastrointestinal disorders) | 79
Vomiting (Gastrointestinal disorders) | 25
Malaise (General disorders) | 26
Nasopharyngitis (Infections and infestations) | 62
Dizziness (Nervous system disorders) | 39
Headache (Nervous system disorders) | 29
Somnolence (Nervous system disorders) | 26
Insomnia (Psychiatric disorders) | 20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2014-11-20): https://cdn.clinicaltrials.gov/large-docs/76/NCT02382276/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-27): https://cdn.clinicaltrials.gov/large-docs/76/NCT02382276/SAP_001.pdf